CLINICAL TRIAL: NCT00403273
Title: Botulinum Toxin A for Painful Total Knee Arthroplasty (TKA): Randomized, Controlled, Triple-blind Study
Brief Title: Safety and Efficacy of Botulinum Toxin A Injection in Patients With Painful Artificial Knee Arthroplasty (TKA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: University of Minnesota (Other); Arthritis Foundation (Other)
Responsible Party: Principal Investigator, jasvinder singh, worker without compensation, Minneapolis Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1-singh
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Results first posted 2016-11-18 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-04

CONDITIONS: Knee Pain
Keywords: Painful Knee Arthroplasty; Botulinum Toxin A; Randomized Controlled Trial; Pain and Function
MeSH Terms: conditions — Pain | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Single Intra-articular Injection of 100 units of Botulinum toxin A in 5 cc of normal saline in the Painful TKA at screening visit
  Interventions: Drug: Botulinum toxin A
- B (Placebo Comparator): Single Intra-articular Injection of 5 cc of normal saline in the Painful TKA at screening visit
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Botulinum toxin A — 100 units of Botulinum toxin A in 5 cc of normal saline in the Painful TKA at screening visit
  Other Names: Botox
  Arms: A
Drug: Normal Saline — Single Intra-articular Injection of 5 cc of normal saline in the Painful TKA at screening visit
  Other Names: saline control
  Arms: B

SUMMARY:
Primary Total Knee joint replacement surgery is highly successful surgery for relieving pain and improving function in patients with disabling arthritis. Unfortunately, like all biomedical devices, prosthesis failure is a complication of knee replacement surgery that leads to disabling pain, stiffness and loss of function. Approximately 1% of the knee replacements fail every year leading to a 20% failure rate over 20 years. The common causes of failure of prosthetic joint are infection, loosening, trauma or wear of the prosthesis. Currently, a revision surgery is the best option for long term pain relief (analgesics or other pain medications are options but are of limited benefit). Surgery may not be feasible in patients due to advancing age, other medical conditions and surgical/technical difficulties or patient's choice. In addition, the results from revision surgery are not as good as the initial knee joint surgery. Therefore, there is a great need for a novel, targeted therapy that provides an option to patients who are unfit, unable, or unwilling to undergo surgery.

In the investigators' recent pilot study, a single injection of Botulinum toxin A (Botox) in painful natural knee, ankle and shoulder joints of patients with various types of arthritis led to significant and durable improvement in pain and function and was safe to use. The investigators propose this 6-month study to compare pain relief, improvement of function and safety of an injection of Botulinum toxin compared to placebo in patients with a painful prosthetic knee joint. Both patients and investigators will be blinded to the treatment assignment to a patient until the study is completed. The investigators will assess the amount and duration of pain relief, improvement in function and short term safety of Botulinum toxin using standard validated measures. Patients will be evaluated at baseline, 2 weeks, 1-, 2-, 3-, 4- and 6-months after a single injection of either placebo or BoNT/A in the hip or knee prosthesis. The six-month follow-up is to assess the duration of meaningful pain relief. If successful, this will offer a new treatment option for patients with a chronically painful knee prosthetic joint, provide more insight into the origin and cause of pain in prosthetic joints and direct future investigations in new directions.

DETAILED DESCRIPTION:
"This 6-month randomized, placebo-controlled, double blind trial will compare a single intra-articular (IA) injection of 100 units of Botulinum Toxin A (BoNT/A) to placebo for improvement in pain, function and quality of life (QOL), and safety in patients with painful total knee arthroplasty (TKA). Patients will be recruited at the Minneapolis VA Medical Center. Patients will be eligible if they are over age 18, have TKA, have pain ≥6/10 on 0-10 numeric rating scale (NRS) and are not candidates for revision surgery.

The primary outcome is: (1) proportion with clinically meaningful change in pain severity (on 0-10 scale) 2 months after IA injection. The choice of 2-month for primary end-point is based on previous observations from open-label case series in painful TKA. Secondary outcomes will be assessed at each efficacy follow-up (FU) visit. The duration of the trial is 6-months to capture the duration of pain relief. Based on other trials of Botulinum toxin, we expect the peak effect between 2-8 weeks and expect the effect to wear off between 2-4 months. Therefore, for all analyses except duration of pain relief, the efficacy time-points (2 wk, 4 wk, 2 month) and possibly 3- or 4-month (depending on duration of pain relief) will be used. Secondary outcomes include: (1) clinically meaningful pain relief (≥2-point or ≥30% decrease) in pain severity (0-10 scale); (2) change in pain severity at 2 months and at all efficacy time-points; (3) percent with Minimal Clinically Important Improvement on Western Ontario MacMaster Arthritis Index (WOMAC) pain and function sub-scales at 2 months and at all efficacy time-points; (4) amount and duration of pain relief; (5) patient and physician global assessment of response at 2 months and at all efficacy time-points; (6) QOL assessed by WOMAC and Short-form 36 (SF-36) scores at 2 months and at all efficacy time-points; (7) change in function by Timed Stands Test (TST) and Timed-up-and-go (TUG) tests at 2 months and at all efficacy time-points; (8) change in dose of analgesics during the study. We will determine time to onset of and duration of pain relief and time to improvement in function. Safety will be assessed by structured interview form for adverse effects, sensory and manual muscle strength testing, and index joint examination for swelling, erythema and tenderness.

At visit #1, after informed consent and screening for inclusion/exclusion criteria, patients will undergo: index joint X-ray, laboratory tests; history, physical examination, index joint pain history, comorbidity and medication history; patient pain assessments, WOMAC and SF-36; and blinded index joint, neurological examination, TST and TUG tests. 50 patients will be randomized to receive either IA BoNT/A 100 units or sterile saline in the index joint. FU phone interviews at 2 and 4-weeks will include pain assessments, WOMAC, patients' global assessment and adverse effects. Interim visits at 2, 3 and 4-months will be identical to visit #1, but will also include patients' and physicians' global assessment and there will be no joint injection. End of study visit at 6 months will be identical to interim visits with the addition of index joint X-ray and laboratory tests.

Main analyses will include patients with unilateral TKAs. Sensitivity analyses will be done by including patients with bilateral knees, accounting for correlatedness of observations. Multiple analysis of variance, mixed model regression analyses and/or generalized estimating equations will be used for analysis of continuous and categorical outcomes respectively. Chi-square tests will be used to compare frequency of adverse events. Analysis will be intention-to-treat.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 years of age or older.
* Written informed consent and written authorization for use or release of health and research study information have been obtained.
* Subject has chronic Prosthetic knee joint pain for more than 3 months.
* Subject has pain 6 or greater on a 10 point Numerical Pain Rating scale
* Ability to follow study instructions and likely to complete all required visits.
* Negative urine pregnancy test on the day of treatment prior to the administration of study medication (for females of childbearing potential). (if applicable)
* Negative infectious etiology workup (joint aspiration, serological parameters such as Erythrocyte Sedimentation Rate (ESR) or C-reactive protein (CRP) and clinical examination).
* Patients who were considered not to be candidates for Prosthetic knee joint revision surgery and have failed traditional treatments including oral pain medications, as determined by referring orthopedic surgeon

Exclusion Criteria:

* Use of aminoglycoside antibiotics, curare-like agents, or other agents that might interfere with neuromuscular function.
* Any medical condition that may put the subject at increased risk with exposure to BOTOX ®including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or known disorders of neuromuscular function
* Females who are pregnant, breast-feeding, or planning a pregnancy during the study or who think that they may be pregnant at the start of the study, or females of childbearing potential who are unable or unwilling to use a reliable form of contraception during the study.
* Know allergy or sensitivity to any of the components in the study medication.
* History of recent or ongoing alcohol or drug abuse.
* Known, uncontrolled systemic disease.
* Concurrent participation in another research study
* Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study.
* Patients whose pain is rated as less than 6 on a 10 point Numerical Pain Rating scale at the screening visit

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jasvinder Singh, MBBS, MPH, Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- Minneapolis VA Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Singh JA, Mahowald ML, Noorbaloochi S. Intraarticular botulinum toxin A for refractory painful total knee arthroplasty: a randomized controlled trial. J Rheumatol. 2010 Nov;37(11):2377-86. doi: 10.3899/jrheum.100336. Epub 2010 Sep 1. PMID 20810509

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 194 TKAs (188 patients) screened, 60 TKAs (54 patients) were recruited in the 6-month study. Main analyses were performed only on 49 TKAs, after excluding bilateral TKAs, to meet the assumption of independence of observations.
Pre-assignment Details: No enrolled participants were excluded from analyses. Main analyses were done for Single TKA per patient, since 6 were bilateral TKAs; sensitivity analyses were done on all, regardless of unilateral or bilateral
Groups:
- Intra-articular Botulinum Toxin: Single Intra-articular Injection of 100 units of Botulinum toxin A in 5 cc of normal saline in the Painful TKA at screening visit
- Intra-articular Placebo: Single Intra-articular Injection of 5 cc of normal saline in the Painful TKA at screening visit
Period: Overall Study
Arm/Group | Intra-articular Botulinum Toxin | Intra-articular Placebo
Started | 25 | 29
Completed | 22 | 25
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 3 | 2
Not completed — Physician Decision | 0 | 1
Not completed — pt. wanted to have a surgical procedure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intra-articular Botulinum Toxin | Intra-articular Placebo | Total
Number analyzed (Participants) | 25 | 29 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (10) | 67 (12) | 67 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 20 | 26 | 46
Race/Ethnicity, Customized [Number; unit: participants]
  caucasian | 24 | 28 | 52
  Non-Caucasian | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Participants With Clinically Meaningful Improvement in Pain Severity (0-10 cm; Higher Score on Pain Scale is Worse)
Description: 2-point reduction in pain Visual Analog Scale (VAS) from baseline to the 2-month follow-up visit, which is considered clinically meaningful Change in Pain Severity; Pain Severity on VAS ranges from 0 (no pain) to 10 (maximum pain)
Time Frame: 2-month post-injection
Population: all with follow-up data, allowing only single TKA per participant
Measure: Number; unit: participants
Arm/Group | Intra-articular Botulinum Toxin | Intra-articular Placebo
Number analyzed (Participants) | 21 | 26
participants | 15 | 9

2. Secondary Outcome: Mean Pain VAS (0-10)
Description: VAS pain score at 2-month post-injection; Pain Severity on VAS ranges from 0 (no pain) to 10 (maximum pain) with higher score indicating worse pain
Time Frame: 2-months post-injection
Population: patients providing pain VAS data at 2-month FU visit
Measure: Mean (Standard Deviation); unit: units on pain VAS scale
Arm/Group | Intra-articular Botulinum Toxin | Intra-articular Placebo
Number analyzed (Participants) | 21 | 26
units on pain VAS scale | 4.4 (2.5) | 5.7 (2.9)

3. Secondary Outcome: Physician Global Assessment of Response to Treatment
Description: Physician global assessed on an ordinal scale with very much improved category as the outcome of interest (compared to all other categories of global assessment as reference category)
Time Frame: 2-month (primary end-point)
Population: 2 patients did not have the outcome assessment; 1 lost to FU
Measure: Number; unit: participants
Arm/Group | Intra-articular Botulinum Toxin | Intra-articular Placebo
Number analyzed (Participants) | 20 | 26
participants | 6 | 0

4. Secondary Outcome: Physical Function Subscale of the WOMAC at 2-months
Description: Physical Function subscale score of the WOMAC at 2-months on a 0 (best physical function) to 100 (worst physical function), with higher score indicating worse physical function
Time Frame: 2-month
Population: people providing data at 2-months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intra-articular Botulinum Toxin | Intra-articular Placebo
Number analyzed (Participants) | 21 | 26
units on a scale | 48.5 (14.1) | 59.7 (17.4)

5. Secondary Outcome: WOMAC Stiffness (0-100)
Description: WOMAC stiffness subscale score on 0-100 scale at 2-month follow-up visit with scores ranging 0 (no joint stiffness) to 100 (worst joint stiffness), with higher score indicating worse joint stiffness
Time Frame: 2-months
Population: patients providing the data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intra-articular Botulinum Toxin | Intra-articular Placebo
Number analyzed (Participants) | 21 | 26
units on a scale | 51.8 (19.1) | 60.4 (16.3)

6. Secondary Outcome: Timed Up-and-go (TUG) Test
Description: Time to get up from a chair, walk 3 meters turn back and sit in the chair in seconds at the 2-month visit (higher number is worse, i.e., taking a longer time to complete the task is worse)
Time Frame: 2-month
Population: patients providing data
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Intra-articular Botulinum Toxin | Intra-articular Placebo
Number analyzed (Participants) | 21 | 26
seconds | 17.2 (18.2) | 9.6 (13.8)

7. Secondary Outcome: QOL: SF-36 Score Physical Functioning Scale, a Generic Health Status Measure
Description: Short Form (SF)-36 physical functioning subscale on 0-100, at 2-month FU visit, as a generic health status measure, with a score ranging from 0 (worst physical functioning) to 100 (best physical functioning), with higher score indicating better physical functioning (higher number is better)
Time Frame: 2-month
Population: patients providing data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intra-articular Botulinum Toxin | Intra-articular Placebo
Number analyzed (Participants) | 21 | 26
units on a scale | 30.7 (21.8) | 23.6 (17.5)

8. Secondary Outcome: Number of Participants With Occurrence of Joint Erythema, Warmth, Swelling or Tenderness
Description: Occurence of any of the above clinical features (erythema, warmth, swelling or tenderness) as a new finding compared to the absence of the same feature at baseline
Time Frame: Upto 6 months
Population: patients providing data
Measure: Number; unit: participants
Arm/Group | Intra-articular Botulinum Toxin | Intra-articular Placebo
Number analyzed (Participants) | 21 | 26
participants | 0 | 0

9. Secondary Outcome: Manual Muscle Strength Testing of Knee Flexion and Extension
Description: Occurence of decrease in strength of knee flexion or extension at any of the follow-up visits, as measured by the Manual muscle strength testing (MMT) with scores ranging 0-5; 0 indicates None: No visible or palpable contraction; 1 indicates Trace: Visible or palpable contraction with no motion; 2 indicates Poor: Full range of motion (ROM) gravity eliminated; 3 indicates Fair: Full ROM against gravity; 4 indicates Good: Full ROM against gravity, moderate resistance; and 5 indicates Normal: Full ROM against gravity, maximal resistance
Time Frame: Upto 6-months
Population: patients providing the data
Measure: Number; unit: participants
Arm/Group | Intra-articular Botulinum Toxin | Intra-articular Placebo
Number analyzed (Participants) | 21 | 26
participants | 0 | 0

10. Secondary Outcome: McGill Affective Dimension
Description: McGill Affective Dimension Score on 0-12 scale at 2-months (higher number is worse)
Time Frame: 2-month
Population: patients providing data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intra-articular Botulinum Toxin | Intra-articular Placebo
Number analyzed (Participants) | 21 | 26
units on a scale | 3.8 (3.1) | 4.8 (3.4)

11. Secondary Outcome: Change in Serum Cytokine (Interleukin 7) Levels at 2-month Post-injection
Description: The change in serum interleukin 7 was defined as the difference between the follow-up (2-month) and the baseline value of serum interleukin 7. We compared the mean change in serum interleukin 7 levels between the WOMAC pain responders vs. the WOMAC pain non-responders.
Time Frame: Baseline to 2-months
Population: This protocol modification was made in the middle of the trial conduct, based on a suggestion on the K-12 application. Therefore, the total number of patients with these data is smaller than the total number of participants.
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- WOMAC Pain Responder: A patient was labeled as a WOMAC Pain responder if the WOMAC pain subscale score decreased by 20 or more on a 0-100 scale from baseline to 2-month follow-up visit.
- WOMAC Pain Non-responder: A patient was labeled as a WOMAC Pain non-responder if the WOMAC pain subscale score decreased by 19 or less on a 0-100 scale from baseline to 2-month follow-up visit.
Arm/Group | WOMAC Pain Responder | WOMAC Pain Non-responder
Number analyzed (Participants) | 12 | 23
pg/ml | 1.07 (1.17) | 0.08 (0.91)
Statistical Analysis 1: Comparison: WOMAC Pain Responder vs WOMAC Pain Non-responder; Test type: Superiority; p = 0.01, t-test, 2 sided — p-value not adjusted for multiple comparisons; the a priori threshold for statistical significance was <0.05

12. Secondary Outcome: McGill Sensory Pain Score
Description: McGill Sensory pain score on 0-33 at 2-month FU visit (higher score is worse)
Time Frame: 2-month
Population: patients providing data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intra-articular Botulinum Toxin | Intra-articular Placebo
Number analyzed (Participants) | 21 | 26
units on a scale | 14.5 (8) | 14.6 (7.5)
Statistical Analysis 1: Comparison: Intra-articular Botulinum Toxin vs Intra-articular Placebo; For primary outcome analysis, we compared the proportion of responders with clinically meaningful change [improvement] in 0-10 VAS Pain, i.e. those with 2-point reduction in 0-10 VAS pain score at 2-mths, in the 2 groups using comparison of proportions. Proportion of responders were also analyzed at all efficacy timepoints using generalized estimating equation (GEE) modeling. We used GEE for between-group comparisons in secondary outcomes at all efficacy endpoints, adjusted for baseline scores; Test type: Superiority or Other; p < 0.05, comparison of proportions — No adjustment for multiple comparisons was made, since we analyzed only one primary outcome. 19 patients per group were needed for 80% power and 24 patients per group for 90% power to detect a difference of 43% in proportion with primary outcome; compare proportion of patients with clinically meaningful change in 0-10 VAS pain (at least 2-point reduction on VAS pain) at 2-mths & all timepoints; comparison of proportions = 0.65 — we hypothesized a greater proportion with meaningful reduction in pain on 0-10 scale in intervention versus placebo group

13. Secondary Outcome: Change in Serum Cytokine (Interleukin 10) Levels at 2-month Post-injection
Description: The change in serum interleukin 10 was defined as the difference between the follow-up (2-month) and the baseline value of serum interleukin 10. We compared the mean change in serum interleukin 10 levels between the WOMAC pain responders vs. the WOMAC pain non-responders.
Time Frame: Baseline to 2-months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | WOMAC Pain Responder | WOMAC Pain Non-responder
Number analyzed (Participants) | 12 | 23
pg/ml | 27.72 (21.56) | 8.51 (20.90)
Statistical Analysis 1: Comparison: WOMAC Pain Responder vs WOMAC Pain Non-responder; Test type: Superiority; p = 0.01, t-test, 2 sided

14. Secondary Outcome: Change in Serum Cytokine (Interleukin 12 p70) Levels at 2-month Post-injection
Description: The change in serum interleukin 12 p70 was defined as the difference between the follow-up (2-month) and the baseline value of serum interleukin 12 p70. We compared the mean change in serum interleukin 12 p70 levels between the WOMAC pain responders vs. the WOMAC pain non-responders.
Time Frame: Baseline to 2-months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | WOMAC Pain Responder | WOMAC Pain Non-responder
Number analyzed (Participants) | 12 | 23
pg/ml | 12.91 (9.60) | 3.36 (8.17)
Statistical Analysis 1: Comparison: WOMAC Pain Responder vs WOMAC Pain Non-responder; Test type: Superiority; p = 0.004, t-test, 2 sided

15. Secondary Outcome: Change in Serum Cytokine (Eotaxin) Levels at 2-month Post-injection
Description: The change in serum Eotaxin was defined as the difference between the follow-up (2-month) and the baseline value of serum Eotaxin. We compared the mean change in serum Eotaxin levels between the WOMAC pain responders vs. the WOMAC pain non-responders.
Time Frame: Baseline to 2-months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | WOMAC Pain Responder | WOMAC Pain Non-responder
Number analyzed (Participants) | 12 | 23
pg/ml | 7.85 (12.28) | -2.03 (13.92)
Statistical Analysis 1: Comparison: WOMAC Pain Responder vs WOMAC Pain Non-responder; Test type: Superiority; p = 0.046, t-test, 2 sided

16. Secondary Outcome: Change in Serum Cytokine (Interferon Gamma) Levels at 2-month Post-injection
Description: The change in serum Interferon Gamma was defined as the difference between the follow-up (2-month) and the baseline value of serum Interferon Gamma. We compared the mean change in serum Interferon Gamma levels between the WOMAC pain responders vs. the WOMAC pain non-responders.
Time Frame: Baseline to 2-months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | WOMAC Pain Responder | WOMAC Pain Non-responder
Number analyzed (Participants) | 12 | 23
pg/ml | 15.61 (13.35) | -1.24 (23.18)
Statistical Analysis 1: Comparison: WOMAC Pain Responder vs WOMAC Pain Non-responder; Test type: Superiority; p = 0.03, t-test, 2 sided

17. Secondary Outcome: Change in Serum Cytokine (Tumor Necrosis Factor Alpha) Levels at 2-month Post-injection
Description: The change in serum tumor necrosis factor alpha was defined as the difference between the follow-up (2-month) and the baseline value of serum tumor necrosis factor alpha. We compared the mean change in serum tumor necrosis factor alpha levels between the WOMAC pain responders vs. the WOMAC pain non-responders.
Time Frame: Baseline to 2-months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | WOMAC Pain Responder | WOMAC Pain Non-responder
Number analyzed (Participants) | 12 | 23
pg/ml | 22.22 (24.65) | 4.46 (21.32)
Statistical Analysis 1: Comparison: WOMAC Pain Responder vs WOMAC Pain Non-responder; Test type: Superiority; p = 0.03, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6-months
Arm/Group | Intra-articular Botulinum Toxin | Intra-articular Placebo
Serious Adverse Events (participants affected / at risk) | 3/23 | 9/26
Other Adverse Events (participants affected / at risk) | 19/23 | 23/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intra-articular Botulinum Toxin (N=23) | Intra-articular Placebo (N=26)
Chest pain/new diagnosis of CAD (Cardiac disorders) | 0 (0) | 3 (3)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Subarachnoid hemorrhage (Cardiac disorders) | 1 (1) | 0 (0)
Atypical chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Seafood allergy (Immune system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis and septic arthritis (Infections and infestations) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Lethargy and decreased appetite (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intra-articular Botulinum Toxin (N=23) | Intra-articular Placebo (N=26)
Accidental injury (Musculoskeletal and connective tissue disorders) | 8 (11) | 6 (7) — Injury as a result of an accident
Pain in the study joint (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2) — Pain reported in the joint that underwent injection
Upper respiratory infections (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 10 (10) — Infections of the upper respiratory tract
Surgical procedure (Surgical and medical procedures) | 3 (3) | 5 (5) — Scheduled surgical procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No